CLINICAL TRIAL: NCT01404325
Title: A 2-arm, Prospective, Randomized, Controlled, Open-label, 12 Month Phase III Trial to Evaluate the Efficacy Regarding Renal Function of Everolimus in Combination With a Centre Specific Standard Immunosuppressive Regimen Consisting of CNI, Purinantagonists and Steroids Versus a Standard Triple Immunosuppressive Regimen in Lung Transplant Recipients.
Brief Title: Efficacy Regarding Renal Function of Everolimus in Combination With Specific Standard Immunosuppressive Regimen Lung Transplant Recipients
Acronym: 4EVERLUNG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ADE36; 2011-001539-21 (EudraCT Number)
Record Dates: First submitted 2011-07-13; First posted 2011-07-28 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-11

CONDITIONS: Lung Transplantation
Keywords: Lung transplantation; everolimus; kidney function; renal function
MeSH Terms: interventions — Standard of Care; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadruple low level IS regimen (Experimental): quadruple immunosuppressive (IS) regimen consisting of everolimus, CNI, MPA and steroids
  Interventions: Drug: Everolimus
- Centre specific triple IS regimen (Experimental): centre specific CNI-based triple drug immunosuppression (IS)
  Interventions: Drug: standard therapy

INTERVENTIONS:
Drug: standard therapy — centre specific CNI-based triple drug immunosuppression
  Arms: Centre specific triple IS regimen
Drug: Everolimus — quadruple immunosuppressive regimen consisting of everolimus, CNI, MPA and steroids
  Other Names: RAD001
  Arms: Quadruple low level IS regimen

SUMMARY:
This trial evaluated the efficacy of an everolimus-based quadruple low immunosuppressive regimen versus a standard immunosuppressive regimen concerning kidney function in lung transplant recipients.

ELIGIBILITY:
Inclusion criteria:

* Adult recipients of de novo cadaveric lung transplants 3-18 months prior to enrollment

Exclusion criteria:

* Patients with thrombocytopenia (platelets <100,000/mm³), with an absolute neutrophil count of <1,500/mm³ or leucopenia (leucocytes <3000/mm³), with anemia with Hb < 8g/dl at time of screening
* Patients with uncontrolled hypercholesterolemia (> 350 mg/dL; > 9.1 mmol/L) or hypertriglyceridemia (> 750 mg/dL; > 8.5 mmol/L) at time of screening
* Patients with a history of malignancy of any organ system, treated or untreated, during the last five years, whether or not there is evidence of local recurrence or metastases, except squamous or basal cell carcinoma of the skin Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Germany (8):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Kneidinger N, Valtin C, Hettich I, Frye BC, Wald A, Wilkens H, Bessa V, Gottlieb J. Five-year Outcome of an Early Everolimus-based Quadruple Immunosuppression in Lung Transplant Recipients: Follow-up of the 4EVERLUNG Study. Transplantation. 2022 Sep 1;106(9):1867-1874. doi: 10.1097/TP.0000000000004095. Epub 2022 Mar 8. PMID 35283454
- [Derived] Gottlieb J, Neurohr C, Muller-Quernheim J, Wirtz H, Sill B, Wilkens H, Bessa V, Knosalla C, Porstner M, Capusan C, Struber M. A randomized trial of everolimus-based quadruple therapy vs standard triple therapy early after lung transplantation. Am J Transplant. 2019 Jun;19(6):1759-1769. doi: 10.1111/ajt.15251. Epub 2019 Feb 5. PMID 30615259

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 232 patients who were de novo lung transplant recipients were planned for enrolling into the study. A total of 130 patients were actually randomized with 67 patients randomized to the quadruple low-level treatment arm and 63 patients randomized to the center-specific triple treatment arm.
Period: Overall Study
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Started | 67 | 63
Completed | 63 | 61
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 2 | 0
Not completed — Graft loss/Retransplantation | 1 | 0
Not completed — non-specified reason | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen | Total
Number analyzed (Participants) | 67 | 63 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (9.5) | 54.2 (9.2) | 54.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Calculated Glomerular Filtration Rate (cGFR) According to Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) at 12 Months
Description: Calculated Glomerular Filtration Rate (cGFR) according to Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) at 12 months The CKD-EPI equation, expressed as a single equation, is GFR = 141 × min(Scr/κ, 1)α × max(Scr/κ, 1)^-1.209 × 0.993Age × 1.018 (if female) × 1.159 (if black), where Scr is serum creatinine, κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/ĸ or 1, and max indicates the maximum of Scr/κ or 1
Time Frame: Month 12
Population: Full Analysis Set multiple imputation (FAS MI) consisted of all patients as randomized that received at least 1 dose of study drug & had a valid baseline assessment of the primary efficacy variable. Missing values was dealt with by multiple imputation (MI)
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
mL/min | 64.5 (16.3) [59.4 to 69.6] | 54.6 (14.3) [49.5 to 59.7]
Statistical Analysis 1: Comparison: Quadruple Low Level IS Regimen vs Centre Specific Triple IS Regimen; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: Calculated Glomerular Filtration Rate (cGFR) According to Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) at Month 1, 3, 6, 9, 12
Description: Calculated Glomerular Filtration Rate (cGFR) according to Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) at Month 1, 3, 6, 9 and 12. The CKD-EPI equation, expressed as a single equation, is GFR = 141 × min(Scr/κ, 1)α × max(Scr/κ, 1)^-1.209 × 0.993Age × 1.018 (if female) × 1.159 (if black), where Scr is serum creatinine, κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/ĸ or 1, and max indicates the maximum of Scr/κ or 1
Time Frame: Month 1, 3, 6, 9, 12
Population: Full Analysis Set (FAS) consisted of all patients as randomized that received at least 1 dose of study drug and had a valid baseline assessment of the primary efficacy variable. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
mL/min
  Month 1 | 73.5 (13.9) | 67.1 (12.4)
  Month 3 | 70.4 (13.3) | 64.3 (12.7)
  Month 6 | 69.2 (15.5) | 63.1 (15.0)
  Month 9 | 69.0 (16.3) | 62.3 (14.8)
  Month 12 | 68.3 (16.3) | 61.2 (14.3)

3. Secondary Outcome: Calculated Glomerular Filtration Rate (cGFR) According to Cystatin C-based Hoek's Formula at Month 1, 3, 6, 9, 12
Description: Calculated Glomerular Filtration Rate (cGFR) according to Cystatin C-based Hoek's formula at Month 1, 3, 6, 9, 12
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
mL/min
  Month 1 | 68.5 (14.6) | 61.8 (12.8)
  Month 3 | 65.7 (15.2) | 60.3 (10.6)
  Month 6 | 63.0 (15.1) | 58.7 (12.2)
  Month 9 | 61.8 (14.1) | 57.7 (12.8)
  Month 12 | 60.8 (14.2) | 57.5 (14.1)

4. Secondary Outcome: Calculated Glomerular Filtration Rate (cGFR) Using Modification of Diet in Renal Disease (MDRD) Formula at Month 1, 3, 6, 9, 12
Description: Calculated Glomerular Filtration Rate (cGFR) Using Modification of Diet in Renal Disease (MDRD) Formula at Month 1, 3, 6, 9, 12 cGFR (in mL/min/1.73 m2) = 186.3*(C-1.154)*(A-0.203)*G*R where C = the serum concentration of creatinine (mg/dL), A = age (years), G = 0.742 when gender is female, otherwise G = 1, R = 1.21 when race is black, otherwise R = 1.
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
mL/min
  Month 1 | 72.0 (13.5) | 65.8 (11.8)
  Month 3 | 68.7 (12.2) | 63.3 (12.3)
  Month 6 | 67.6 (14.1) | 62.3 (15.0)
  Month 9 | 67.4 (14.9) | 61.7 (15.1)
  Month 12 | 67.0 (14.8) | 60.5 (14.4)

5. Secondary Outcome: Calculated Glomerular Filtration Rate (cGFR) According to Cockcroft-Gault at Month 1, 3, 6, 9, 12
Description: Calculated Glomerular Filtration Rate (cGFR) according to Cockcroft-Gault at Month 1, 3, 6, 9, 12 For men: GFR=(140-Age) x Body weight (kg) / 72 x Serum Creatinine (mg/dl) For women: GFR=0.85 (140 -Age) x Body weight(kg)/ 72 x Serum Creatinine (mg/dl)
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
mL/min
  Month 1 | 78.6 (19.2) | 72.1 (14.9)
  Month 3 | 76.1 (17.6) | 70.1 (16.0)
  Month 6 | 76.2 (19.3) | 69.1 (17.5)
  Month 9 | 76.2 (20.1) | 69.0 (18.2)
  Month 12 | 76.2 (20.6) | 68.4 (17.8)

6. Secondary Outcome: Incidence of Patients Experiencing a Decline in GFR of < 10, 10-15, 15-20, 20-25 and > 25 mL/Min From Baseline to Month 6 and 12.
Description: Incidence of patients experiencing a decline in GFR of < 10, 10-15, 15-20, 20-25 and > 25 mL/min from Baseline to Month 6 and 12calculated by the CKD-EPI method. Participants are counted in each decline level observed for that participant; this means participants may be counted in more than 1 decline level.
Time Frame: Baseline, Month 6, Month 12
Population: as for outcome 2
Measure: Number; unit: incidences
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
incidences
  Up to Month 6: < 10 mL/min | 28 | 44
  Up to Month 6: 10 - < 15 mL/min | 9 | 18
  Up to Month 6: 15 - < 20 mL/min | 6 | 11
  Up to Month 6: 20 - < 25 mL/min | 2 | 7
  Up to Month 6: > 25 mL/min | 3 | 7
  Up to Month 12: < 10 mL/min | 36 | 53
  Up to Month 12: 10 - < 15 mL/min | 10 | 27
  Up to Month 12: 15 - < 20 mL/min | 8 | 18
  Up to Month 12: 20 - < 25 mL/min | 8 | 9
  Up to Month 12: > 25 mL/min | 7 | 9

7. Secondary Outcome: Incidence of Renal Replacement Therapy at Month 6 and Month 12
Description: Incidence of renal replacement therapy at Month 6 and Month 12: There were no incidences in either group where renal replacement therapy was required
Time Frame: Month 6, Month 12
Population: as for outcome 2
Measure: Number; unit: incidences
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
incidences
  up to Month 6 | 0 | 0
  up to Month 12 | 0 | 0

8. Secondary Outcome: Time to Renal Replacement Therapy at Month 6 and Month 12
Description: Time to renal replacement therapy at Month 6 and Month 12: There were no incidences in either group where renal replacement therapy was required
Time Frame: Month 6, Month 12
Population: Full Analysis Set (FAS) consisted of all patients as randomized that received at least 1 dose of study drug and had a valid baseline assessment of the primary efficacy variable. The outcome could not be analyzed because there were no incidences of renal replacement therapy
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Incidence of Acute Rejection Episodes at Month 6 and Month 12
Description: Incidence of acute rejection episodes at Month 6 and Month 12. This table counts multiple occurrences of rejection in the same patient as different incidents. Every incident is associated with both an A and a B classification.
  Classification A: Acute Rejection Grade 0 - none, Grade 1-minimal, Grade 2- mild, Grade 3-moderate, Grade 4-Severe; Classification B: Airway Inflammation-Grade 0-none, Grade 1R-low grade, Grade 2R-high grade, Grade X-ungradeable
Time Frame: Month 6, Month 12
Population: as for outcome 2
Measure: Number; unit: incidences
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
incidences
  Up to 6 months: Classification A | 11 | 13
  Up to 6 months: Classification B | 11 | 13
  6 to 12 months: Classification A | 10 | 9
  6 to 12 months: Classification B | 10 | 9

10. Secondary Outcome: Incidence of Graft Loss/Re-transplantation at Month 6 and Month 12
Description: Incidence of graft loss/re-transplantation at Month 6 and Month 12
Time Frame: Month 6, Month 12
Population: as for outcome 2
Measure: Number; unit: incidences
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
incidences
  Month 6 | 0 | 0
  Month 12 | 1 | 1

11. Secondary Outcome: Incidence of Bronchiolitis Obliterans Syndrome (BOS) at Month 6 and Month 12
Description: Incidence of Bronchiolitis obliterans syndrome (BOS) at Month 6 and Month 12 BOS 0 is FEV1 > 90% of baseline and FEF25-75% > 75% of baseline; BOS 0-p is FEV1 81-90% of baseline and/or FEF25-75% ≤ 75% of baseline; BOS 1 is FEV1 66-80% of baseline; BOS 2 is FEV1 51-65% of baseline; BOS 3 is FEV1 ≤ 50% of baseline
Time Frame: Month 6, Month 12
Population: as for outcome 2
Measure: Number; unit: incidences
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
incidences
  Month 6 - Total (all grades) | 66 | 61
  Month 6 - BOS 0 | 36 | 40
  Month 6 - BOS 0p | 26 | 14
  Month 6 - BOS 1 | 3 | 5
  Month 6 - BOS 2 | 1 | 0
  Month 6 - BOS 3 | 0 | 2
  Month 6 - BOS (>/=1) | 4 | 7
  Month 12 - Total (all grades) | 66 | 61
  Month 12 - BOS 0 | 35 | 38
  Month 12 - BOS 0p | 26 | 14
  Month 12 - BOS 1 | 3 | 5
  Month 12 - BOS 2 | 1 | 1
  Month 12 - BOS 3 | 1 | 3
  Month 12 - BOS (>/=1) | 5 | 9

12. Secondary Outcome: Incidence of Death at Month 6 and Month 12
Description: Incidence of death at Month 6 and Month 12
Time Frame: Month 6, Month 12
Population: Safety Set consisted of all patients that received at least 1 dose of study drug and had at least 1 post-baseline safety assessment. Patients were analyzed according to treatment received. Of note, the statement that a patient had no AEs also constituted a safety assessment.
Measure: Number; unit: incidences
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
incidences
  Month 6 | 0 | 0
  Month 12 | 3 | 1

13. Secondary Outcome: Quality of Life (QoL, SF36) at Month 6 and Month 12
Description: Quality of Life (QoL, SF36) at Month 6 and Month 12 Scores can range from a minimum of 0 (maximum disability) to a maximum of 100 (no disability).
Time Frame: Month 6, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
scores on a scale
  Month 6: Physical component summary score | 46.9 (7.6) | 48.9 (7.3)
  Month 6: Mental component summary score | 51.5 (10.8) | 52.6 (8.1)
  Month 6: Physical functioning | 78.8 (20.9) | 84.1 (16.8)
  Month 6: Role-Physical | 71.1 (23.2) | 77.1 (24.2)
  Month 6: Bodily pain | 76.4 (27.9) | 81.3 (23.4)
  Month 6: General health perception | 65.4 (19.2) | 70.6 (19.9)
  Month 6: Vitality | 67.4 (18.0) | 70.0 (14.6)
  Month 6:Social functioning | 84.1 (22.6) | 88.9 (17.6)
  Month 6: Role-Emotional | 84.7 (22.4) | 84.8 (17.9)
  Month 6: Mental health | 78.5 (17.2) | 81.0 (12.8)
  Month 12: Physical component summary score | 47.2 (8.8) | 47.7 (7.1)
  Month 12: Mental component summary score | 49.7 (11.8) | 53.8 (9.1)
  Month 12: Physical functioning | 77.4 (21.8) | 82.5 (20.0)
  Month 12: Role-Physical | 68.3 (26.8) | 78.0 (22.9)
  Month 12: Bodily Pain | 76.8 (27.0) | 80.1 (22.7)
  Month 12: General health perception | 66.7 (17.3) | 65.8 (20.3)
  Month 12: Vitality | 65.7 (19.4) | 69.9 (17.5)
  Month 12: Social functioning | 82.3 (23.0) | 90.5 (16.1)
  Month 12: Role-Emotional | 79.4 (27.3) | 86.2 (20.5)
  Month 12: Mental health | 75.4 (18.2) | 81.8 (14.8)

14. Secondary Outcome: Exercise Capacity 6-Minute Walk Test(6MWT) at Month 6 and Month 12
Description: Exercise capacity (6MWT) at Month 6 and Month 12 Measured by the Borg Scale. THE BORG SCALE 0 is Nothing at all, 0.5 is Very, very slight (just noticeable); 1 is Very slight, 2 is Slight (light); 3 is Moderate; 4 is Somewhat severe; 5 is Severe (heavy), 7 is Very severe, 10 is Very, very severe (maximal)The higher the Borg score implies increased shortness of breath and/or increased fatigue.
Time Frame: Month 6, Month 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
Scores on a scale
  Month 6-Borg score - Before start of test | 0.47 (0.78) | 0.39 (0.77)
  Month 6-Borg score - At end of test | 1.75 (1.58) | 1.64 (1.31)
  Month 12-Borg score - Before start of test | 0.38 (0.94) | 0.42 (0.79)
  Month 12-Borg score - At end of test | 2.08 (1.58) | 2.06 (1.85)

15. Secondary Outcome: Incidence of Treated Arterial Hypertension up to Month 12
Description: Incidence of treated of arterial hypertension up to Month 12
Time Frame: up to Month 12
Population: as for outcome 2
Measure: Number; unit: incidences
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
incidences
  Month 1 | 2 | 1
  Month 3 | 2 | 1
  Month 6 | 2 | 1
  Month 9 | 3 | 1
  Month 12 | 4 | 1

16. Secondary Outcome: Incidence of Diabetes Mellitus up to Month 12
Description: Incidence of Diabetes Mellitus up to Month 12
Time Frame: up to Month 12
Population: as for outcome 2
Measure: Number; unit: incidences
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
incidences
  Month 1 | 0 | 0
  Month 3 | 0 | 0
  Month 6 | 0 | 1
  Month 9 | 1 | 1
  Month 12 | 1 | 1

17. Secondary Outcome: Trough Levels of Everolimus at Month 1, 3, 6, 9, 12
Description: Trough levels of everolimus at Month 1, 3, 6, 9, 12
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Quadruple Low Level IS Regimen
Number analyzed (Participants) | 67
ng/mL
  Month 1: number analyzed (Participants) | 66
  Month 1 | 4.2 (1.4)
  Month 3: number analyzed (Participants) | 61
  Month 3 | 4.4 (1.2)
  Month 6: number analyzed (Participants) | 58
  Month 6 | 4.1 (1.2)
  Month 9: number analyzed (Participants) | 52
  Month 9 | 4.5 (1.6)
  Month 12: number analyzed (Participants) | 50
  Month 12 | 4.3 (1.1)

18. Secondary Outcome: Adherence to Target Ranges of Everolimus at Month 1, 3, 6, 9, 12
Description: Adherence to target ranges of everolimus at Month 1, 3, 6, 9, 12
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 12
Measure: Number; unit: participant adherence
Arm/Group | Quadruple Low Level IS Regimen
Number analyzed (Participants) | 67
participant adherence
  Month 1 Below Target Range | 10 (1.4)
  Month 1 Within Target Range | 42 (1.2)
  Month 1 Above Target Range | 14 (1.2)
  Month 3 Below Target Range | 5 (1.6)
  Month 3 Within Target Range | 41 (1.1)
  Month 3 Above Target Range | 15
  Month 6 Below Target Range | 7
  Month 6 Within Target Range | 39
  Month 6 Above Target Range | 12
  Month 9 Below Target Range | 5
  Month 9 Within Target Range | 34
  Month 9 Above Target Range | 13
  Month 12 Below Target Range | 3
  Month 12 Within Target Range | 38
  Month 12 Above Target Range | 9

19. Secondary Outcome: Trough Levels of Cyclosporine A (CsA) at Month 1, 3, 6, 9, 12
Description: Trough levels of Cyclosporine A (CsA) at Month 1, 3, 6, 9, 12
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
ng/mL
  Month 1: number analyzed (Participants) | 21 | 16
  Month 1 | 61 (21.83) | 106 (21.25)
  Month 3: number analyzed (Participants) | 20 | 14
  Month 3 | 59.65 (20.43) | 109 (24.95)
  Month 6: number analyzed (Participants) | 20 | 14
  Month 6 | 58.50 (12.84) | 103 (32.95)
  Month 9: number analyzed (Participants) | 17 | 13
  Month 9 | 57.59 (23.26) | 107 (29.13)
  Month 12: number analyzed (Participants) | 21 | 13
  Month 12 | 69.33 (48.41) | 108 (27.82)

20. Secondary Outcome: Adherence to Target Ranges of Cyclosporine A (CsA) at Month 1, 3, 6, 9, 12
Description: Adherence to target ranges of Cyclosporine A (CsA) at Month 1, 3, 6, 9, 12
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 12
Measure: Number; unit: participant adherence
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
participant adherence
  Month 1 Below Target Range | 0 (21.83) | 8 (21.25)
  Month 1 Within Target Range | 18 (20.43) | 8 (24.95)
  Month 1 Above Target Range | 3 (12.84) | 0 (32.95)
  Month 3 Below Target Range | 0 (23.26) | 4 (29.13)
  Month 3 Within Target Range | 18 (48.41) | 10 (27.82)
  Month 3 Above Target Range | 2 | 0
  Month 6 Below Target Range | 0 | 6
  Month 6 Within Target Range | 18 | 8
  Month 6 Above Target Range | 2 | 0
  Month 9 Below Target Range | 0 | 4
  Month 9 Within Target Range | 16 | 9
  Month 9 Above Target Range | 1 | 0
  Month 12 Below Target Range | 0 | 3
  Month 12 Within Target Range | 16 | 10
  Month 12 Above Target Range | 5 | 0

21. Secondary Outcome: Trough Levels of Tacrolimus at Month 1, 3, 6, 9, 12
Description: Trough levels of Tacrolimus at Month 1, 3, 6, 9, 12
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
ng/mL
  Month 1: number analyzed (Participants) | 44 | 45
  Month 1 | 5.07 (1.80) | 10.44 (2.73)
  Month 3: number analyzed (Participants) | 44 | 47
  Month 3 | 5.18 (2.02) | 10.53 (2.88)
  Month 6: number analyzed (Participants) | 40 | 46
  Month 6 | 4.70 (1.98) | 10.09 (3.37)
  Month 9: number analyzed (Participants) | 38 | 46
  Month 9 | 5.78 (4.18) | 10.67 (3.44)
  Month 12: number analyzed (Participants) | 41 | 47
  Month 12 | 5.19 (2.36) | 9.66 (3.01)

22. Secondary Outcome: Adherence to Target Ranges of Tacrolimus at Month 1, 3, 6, 9, 12
Description: Adherence to target ranges of Tacrolimus at Month 1, 3, 6, 9, 12
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 12
Measure: Number; unit: participant adherence
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
participant adherence
  Month 1 Below Target Range | 3 (21.83) | 0 (21.25)
  Month 1 Within Target Range | 24 (20.43) | 45 (24.95)
  Month 1 Above Target Range | 17 (12.84) | 0 (32.95)
  Month 3 Below Target Range | 3 (23.26) | 0 (29.13)
  Month 3 Within Target Range | 23 (48.41) | 47 (27.82)
  Month 3 Above Target Range | 18 | 0
  Month 6 Below Target Range | 5 | 1
  Month 6 Within Target Range | 23 | 45
  Month 6 Above Target Range | 12 | 0
  Month 9 Below Target Range | 2 | 0
  Month 9 Within Target Range | 18 | 46
  Month 9 Above Target Range | 18 | 0
  Month 12 Below Target Range | 3 | 0
  Month 12 Within Target Range | 23 | 47
  Month 12 Above Target Range | 15 | 0

23. Secondary Outcome: Incidence of Bacterial, Viral, and Fungal Infections at Month 12
Description: Incidence of bacterial, viral, and fungal infections at Month 12
Time Frame: Month 12
Population: as for outcome 12
Measure: Number; unit: incidences
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
incidences
  Bacterial infections | 3 | 4
  Viral infections | 14 | 20
  Fungal infections | 3 | 0

24. Secondary Outcome: Triglyceride Levels at Month 1, 3, 6, 9, 12
Description: Triglyceride levels at Month 1, 3, 6, 9, 12
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
mmol/L
  Month 1: number analyzed (Participants) | 66 | 60
  Month 1 | 2.6 (1.4) | 2.0 (0.9)
  Month 3: number analyzed (Participants) | 65 | 60
  Month 3 | 2.7 (1.3) | 2.1 (1.0)
  Month 6: number analyzed (Participants) | 60 | 60
  Month 6 | 2.6 (1.2) | 2.0 (1.1)
  Month 9: number analyzed (Participants) | 55 | 59
  Month 9 | 2.7 (1.3) | 2.0 (1.0)
  Month 12: number analyzed (Participants) | 63 | 60
  Month 12 | 2.7 (1.5) | 2.1 (0.9)

25. Secondary Outcome: Total Cholesterol Levels at Month 1, 3, 6, 9, 12
Description: Total Cholesterol levels at Month 1, 3, 6, 9, 12
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
mmol/L
  Month 1: number analyzed (Participants) | 64 | 60
  Month 1 | 0.8 (0.8) | -0.2 (0.7)
  Month 3: number analyzed (Participants) | 63 | 60
  Month 3 | 1.0 (0.8) | -0.1 (0.9)
  Month 6: number analyzed (Participants) | 59 | 60
  Month 6 | 1.1 (0.9) | -0.2 (0.8)
  Month 9: number analyzed (Participants) | 54 | 59
  Month 9 | 1.1 (0.9) | -0.1 (0.9)
  Month 12: number analyzed (Participants) | 61 | 60
  Month 12 | 0.8 (1.1) | -0.1 (0.8)

26. Secondary Outcome: Low-Density Lipoprotein (LDL)Cholesterol Levels at Month 1, 3, 6, 9, 12
Description: LDL Cholesterol levels at Month 1, 3, 6, 9, 12
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
mmol/L
  Month 1: number analyzed (Participants) | 63 | 57
  Month 1 | 0.4 (0.8) | 0.0 (0.5)
  Month 3: number analyzed (Participants) | 62 | 58
  Month 3 | 0.6 (0.7) | -0.0 (0.6)
  Month 6: number analyzed (Participants) | 58 | 57
  Month 6 | 0.7 (0.8) | -0.0 (0.6)
  Month 9: number analyzed (Participants) | 53 | 56
  Month 9 | 0.8 (0.8) | 0.1 (0.7)
  Month 12: number analyzed (Participants) | 57 | 57
  Month 12 | 0.5 (0.9) | 0.1 (0.6)

27. Secondary Outcome: High-Density Lipoprotein (HDL)Cholesterol Levels at Month 1, 3, 6, 9, 12
Description: HDL Cholesterol levels at Month 1, 3, 6, 9, 12
Time Frame: Month 1, 3, 6, 9, 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Number analyzed (Participants) | 67 | 63
mmol/L
  Month 1: number analyzed (Participants) | 65 | 59
  Month 1 | 0.1 (0.3) | -0.1 (0.3)
  Month 3: number analyzed (Participants) | 64 | 59
  Month 3 | 0.1 (0.3) | -0.0 (0.4)
  Month 6: number analyzed (Participants) | 60 | 59
  Month 6 | 0.1 (0.4) | -0.0 (0.4)
  Month 9: number analyzed (Participants) | 55 | 58
  Month 9 | 0.0 (0.4) | -0.0 (0.4)
  Month 12: number analyzed (Participants) | 59 | 59
  Month 12 | 0.0 (0.5) | -0.0 (0.4)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until 12 months.
Arm/Group | Quadruple Low Level IS Regimen | Centre Specific Triple IS Regimen
Serious Adverse Events (participants affected / at risk) | 29/67 | 22/63
Other Adverse Events (participants affected / at risk) | 62/67 | 58/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Quadruple Low Level IS Regimen (N=67) | Centre Specific Triple IS Regimen (N=63)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0
COR PULMONALE (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 2 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1
HYDROCELE (Congenital, familial and genetic disorders) | 1 | 0
RETINAL DETACHMENT (Eye disorders) | 1 | 0
RETINAL VEIN OCCLUSION (Eye disorders) | 0 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 2
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
HAEMORRHAGIC EROSIVE GASTRITIS (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 1
CHEST PAIN (General disorders) | 3 | 0
CHILLS (General disorders) | 1 | 0
HERNIA (General disorders) | 0 | 2
INFLAMMATION (General disorders) | 0 | 1
LOCAL SWELLING (General disorders) | 0 | 1
LOCALISED OEDEMA (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 3 | 0
PERIPHERAL SWELLING (General disorders) | 1 | 0
PYREXIA (General disorders) | 4 | 3
LUNG TRANSPLANT REJECTION (Immune system disorders) | 5 | 0
ATYPICAL PNEUMONIA (Infections and infestations) | 0 | 1
BRONCHITIS (Infections and infestations) | 2 | 1
BRONCHITIS BACTERIAL (Infections and infestations) | 1 | 0
BRONCHITIS VIRAL (Infections and infestations) | 0 | 1
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 | 4
GASTROENTERITIS (Infections and infestations) | 1 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 1
INFECTION (Infections and infestations) | 3 | 2
LUNG INFECTION (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 3 | 3
PNEUMONIA VIRAL (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 1 | 0
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 3
SUPERINFECTION BACTERIAL (Infections and infestations) | 0 | 1
TRACHEOBRONCHITIS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
UROSEPSIS (Infections and infestations) | 1 | 0
COMPLICATIONS OF TRANSPLANTED LUNG (Injury, poisoning and procedural complications) | 1 | 0
MATERNAL EXPOSURE DURING PREGNANCY (Injury, poisoning and procedural complications) | 0 | 1
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 | 0
FORCED EXPIRATORY VOLUME DECREASED (Investigations) | 9 | 5
IMMUNOSUPPRESSANT DRUG LEVEL INCREASED (Investigations) | 0 | 1
PULMONARY FUNCTION TEST DECREASED (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
PSEUDARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0
PARAPARESIS (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 1 | 0
TREMOR (Nervous system disorders) | 1 | 0
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 1
URGE INCONTINENCE (Renal and urinary disorders) | 1 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 2 | 0
BRONCHOSTENOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 4
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
IDIOPATHIC PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 3 | 0
OBLITERATIVE BRONCHIOLITIS (Respiratory, thoracic and mediastinal disorders) | 3 | 1
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 2
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0
LYMPHOCELE (Vascular disorders) | 0 | 1
LYMPHORRHOEA (Vascular disorders) | 0 | 1
PERIPHERAL VENOUS DISEASE (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quadruple Low Level IS Regimen (N=67) | Centre Specific Triple IS Regimen (N=63)
ANAEMIA (Blood and lymphatic system disorders) | 6 | 3
LEUKOPENIA (Blood and lymphatic system disorders) | 15 | 19
DIARRHOEA (Gastrointestinal disorders) | 9 | 10
NAUSEA (Gastrointestinal disorders) | 9 | 10
VOMITING (Gastrointestinal disorders) | 5 | 4
CHEST PAIN (General disorders) | 2 | 5
OEDEMA PERIPHERAL (General disorders) | 19 | 10
PYREXIA (General disorders) | 1 | 5
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 10 | 11
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 4
NASOPHARYNGITIS (Infections and infestations) | 17 | 17
RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 | 7
URINARY TRACT INFECTION (Infections and infestations) | 4 | 2
COMPLICATIONS OF TRANSPLANTED LUNG (Injury, poisoning and procedural complications) | 0 | 4
BRONCHOALVEOLAR LAVAGE ABNORMAL (Investigations) | 3 | 6
C-REACTIVE PROTEIN INCREASED (Investigations) | 2 | 4
FORCED EXPIRATORY VOLUME DECREASED (Investigations) | 7 | 8
PULMONARY FUNCTION TEST DECREASED (Investigations) | 6 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 5
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 | 5
HEADACHE (Nervous system disorders) | 8 | 9
MIGRAINE (Nervous system disorders) | 3 | 4
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 | 7
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 4
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 5
ACNE (Skin and subcutaneous tissue disorders) | 12 | 1
HYPERTENSION (Vascular disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single- site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.